CLINICAL TRIAL: NCT06376968
Title: Prospective, Multicentre, Randomized, Controlled, Cross-over Study on the Safety and Performance of the Biologic Fusion Option of DialogiQ Compared to Haemodialysis Without Biologic Fusion in Hypotension Prone Patients on Maintenance Haemodialysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: B.Braun Avitum AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BA-G-H-1604
Record Dates: First submitted 2024-04-16; First posted 2024-04-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BioLogic Fusion followed by standard dialysis (Experimental): Patients will be dialysed first with the BioLogic Fusion feature activated and then switched to standard dialysis with the BioLogic Fusion feature de-activated
  Interventions: Device: BioLogic Fusion
- Standard dialysis followed by BioLogic Fusion (Experimental): Patients will be dialysed first with standard dialysis with the BioLogic Fusion feature de-activated and then switched to the BioLogic Fusion feature activated
  Interventions: Device: BioLogic Fusion

INTERVENTIONS:
Device: BioLogic Fusion — Dialysis conducted with Dialog iQ dialysis machine either using the BioLogic Fusion option or not using it. This is only a biologic feedback system using blood pressure and residual blood volume as parameters to predict potential hypotensive episodes. If switched off, standard dialysis treatment happens, if switched on, the system tries to predict and prevent hypotensive episodes.

SUMMARY:
The goal of this prospective, randomized, controlled, cross-over, multicentric study is to demonstrate the safety of bioLogic Fusion in patients on chronic haemodialysis or hemodiafiltration prone to hypotensive episodes. The main question it aims to answer is:

• Which is the number and percentage of individual sessions with reached prescribed post-dialysis body weight in the prescribed treatment time in each single session in hypotensive-prone patients on high-flux haemodialysis or hemodiafiltration within each patient with treatments performed with DialogiQ with (treatment A) or without (treatment B) the bioLogic Fusion option activated? Participants will in addition to their routine dialysis treatment undergo 2 physical examinations and regularly answer questionnaires.

A crossover design is used to compare treatments with or without the BioLogic Fusion function activated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 years of age
* Chronic bicarbonate standard high-flux haemodialysis or hemodiafiltration for at least 3 months
* Dialysis frequency 3 x per week
* Dialysis duration per session ≥ 4h
* Patient on chronic haemodialysis or hemodiafiltration prone to hypotensive episodes
* No residual renal function (definition: ≤100 ml urine/day) - changed to "No to minimal residual renal function (definition: ≤ 300 ml/day)" with Amendment 1 (CIP version 6)
* Stable dry body weight for at least 4 weeks
* Subjects who are willing to give a voluntary consent to participate in the study

Exclusion Criteria:

* Simultaneous participation in another interventional clinical trial (drugs or medical devices studies)
* Vascular access insufficiency (mean blood flow <200ml/min)
* Patients treated with dialysis profiles: sodium profile, Ultrafiltration (UF) profile, and temperature profile - changed to: " Patients treated with dialysis profiles during the 9 prescreening visits: sodium profile, UF profile, and temperature profile. However, patients on sodium, ultrafiltration or temperature profiling expected to reduce intradialytic hypotensive episodes can be evaluated for enrollment when their frequency of sessions complicated by hypotension demonstrate the lack of efficacy of the applied profiles" with Amendment 1 (CIP version 6)
* Use of the BioLogic fusion function during the last 9 dialysis sessions recorded at the site (retrospective screening period)
* Pregnant or nursing women. Women of childbearing potential must agree to avoid pregnancy during the study period
* Factors which may interfere with full participation in the trial
* Any contra-indication to haemodialysis treatment per se, as described in the Instructions for Use (IFU)
* Any serious medical condition or disability, which in the opinion of the investigator limits the life expectancy and would preclude completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Post-dialysis body weight | 12 weeks
  percentage of sessions with reached prescribed post-dialysis body weight

CONTACTS AND LOCATIONS:
Overall Officials: Annalisa Zucchelli, MD, Principal Investigator — University Hospital Bologna
Locations (1):
- Policlinico S. Orsola - Malpighi - UOC Nefrologia, Dialisi e Ipertensione, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No